CLINICAL TRIAL: NCT03854487
Title: Effect of Mirror Therapy on Unilateral Neglect for Patients After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Tung Wah Hospital (Other); Guangdong 999 Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BQ46L
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: The Effects of Mirror Therapy on Patients With Unilateral Neglect After Stroke
Keywords: stroke; unilateral neglect; mirror therapy; mirror visual feedback
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mirror therapy (Experimental)
  Interventions: Behavioral: Mirror therapy
- Sham mirror (Sham Comparator)
  Interventions: Behavioral: Sham mirror
- Covered mirror (Active Comparator)
  Interventions: Behavioral: Covered mirror

INTERVENTIONS:
Behavioral: Mirror therapy — A mirror is placed at the midsagittal plane of the patient. The patients in the mirror therapy group watched the mirror illusion of the non-affected arm in the mirror and moved together with the affected arm. The treatment programme for all groups consisted of 12 sessions (4 per week for 3 weeks), each lasting for 30 minutes. The movement practice involved 5 table-top tasks and the patient was instructed to perform as many trials as possible in each session with a maximum of 30 trials per task, giving a total of 150 trials per session. Treatment activities are graded according to the severity of the patient's upper extremity impairment.
  Arms: Mirror therapy
Behavioral: Sham mirror — A transparent glass wall is placed at the midsagittal plane of the patient. The patients in the sham mirror group watched the movements of the affected arm through the transparent glass wall and moved together with the non-affected arm. The treatment programme for all groups consisted of 12 sessions (4 per week for 3 weeks), each lasting for 30 minutes. The movement practice involved 5 table-top tasks and the patient was instructed to perform as many trials as possible in each session with a maximum of 30 trials per task, giving a total of 150 trials per session. Treatment activities are graded according to the severity of the patient's upper extremity impairment.
  Arms: Sham mirror
Behavioral: Covered mirror — A covered mirror is placed at the midsagittal plane of the patient. The patients in the control group watched the movements of the non-affected arm and moved together with the affected arm behind the covered mirror. The treatment programme for all groups consisted of 12 sessions (4 per week for 3 weeks), each lasting for 30 minutes. The movement practice involved 5 table-top tasks and the patient was instructed to perform as many trials as possible in each session with a maximum of 30 trials per task, giving a total of 150 trials per session. Treatment activities are graded according to the severity of the patient's upper extremity impairment.
  Arms: Covered mirror

SUMMARY:
This is a single-blinded randomized controlled trial to investigate the effects of mirror therapy (MT), with reference to sham mirror (a glass wall) and control (a covered mirror), in reducing unilateral neglect for patients with stroke in 2 centres.

DETAILED DESCRIPTION:
Twenty-one subacute inpatients with left unilateral neglect after right-hemispheric stroke, recruited from 2 hospitals - Hong Kong and Guangzhou, in 1 and a half years, were randomly assigned to three groups; mirror therapy, sham therapy (in the form of a transparent glass wall), and control (covered mirror). The treatment programme for all groups consisted of 12 sessions (4 per week for 3 weeks) movement practice for the hemiplegic arm involved 5 table-top tasks graded according to the severity of patients' arm impairments. Blinded assessments were administered at baseline, 3-week postintervention, and 3-week follow-up upon completion of training.

ELIGIBILITY:
Inclusion Criteria:

* ischemic or hemorrhagic stroke, confirmed by medical diagnoses compatible with a unilateral right lesion involvement (i.e. left hemiplegic), exhibited left visual field inattention or unilateral neglect by obtaining a total score of star cancellation subtest in the conventional battery of the Behavioural Inattention Test ≤ 51 (out of 54);
* stroke with onset of neurological condition ≤ 6 months previously;
* have normal or corrected-to-normal visual acuity better than 20/60 (6/18) in the better eye;
* with hemiplegic upper extremity functional levels 3-7 as rated by Functional Test for the Hemiplegic Upper Extremity and is able to move against gravity;
* ability to understand and follow simple verbal instructions, with Mini-mental State Examination ≥ 21;
* ability to participate in a therapy session lasting at least 30 minutes;
* consent to participant in the study

Exclusion Criteria:

* prior neurological or psychiatric disorders;
* severe spasticity (Modified Ashworth Scale >3) over paretic arm;
* history of recent Botox injection or acupuncture to the paretic arm within the past three months;
* participation in another clinical study elsewhere apart from the study site during recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, Female
Enrollment: 21 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Unilateral neglect | Change of baseline to 3-week and to follow-up at 6-week
  Behavioural Inattention Test
Allocentric and egocentric neglect | Change of baseline to 3-week and to follow-up at 6-week
  Gap Detection Test
Functional performance related to unilateral neglect | Change of baseline to 3-week and to follow-up at 6-week
  Catherine Bergego Scale

SECONDARY OUTCOMES:
Upper limb functions | Change of baseline to 3-week and to follow-up at 6-week
  Fugl-Meyer assessment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Longley V, Hazelton C, Heal C, Pollock A, Woodward-Nutt K, Mitchell C, Pobric G, Vail A, Bowen A. Non-pharmacological interventions for spatial neglect or inattention following stroke and other non-progressive brain injury. Cochrane Database Syst Rev. 2021 Jul 1;7(7):CD003586. doi: 10.1002/14651858.CD003586.pub4. PMID 34196963